CLINICAL TRIAL: NCT01285180
Title: Daxas in COPD Therapy
Brief Title: Quality of Life in Daxas-treated Patients Older Than 18 Years With Severe COPD
Acronym: DINO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-2455-402-DE; U1111-1136-8860 (Registry Identifier: WHO)
Record Dates: First submitted 2011-01-21; First posted 2011-01-27 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Severe COPD
Keywords: COPD; Quality of life; sociodemographic data; cost-of-illness data; roflumilast; Daxas
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DINO
  Interventions: Drug: Daxas

INTERVENTIONS:
Drug: Daxas — 500 microgram, oral, once daily as add-on therapy to existing therapy

SUMMARY:
Daxas (roflumilast) is the first oral anti-inflammatory phosphodiesterase inhibitor (PDE-4) for patients with severe chronic obstructive pulmonary disease (COPD) experiencing chronic cough and sputum and with a history of exacerbations as add-on to bronchodilator treatment. With its mode of action Daxas can reduce exacerbations rates and improve lung function parameters which may result in a better health-related quality of life and an improved long-term management of COPD.

The aim of this non-interventional study is to evaluate data on quality of life in COPD patients in Germany in a real life medical setting. Evaluation is based on two COPD specific questionnaires to assess the patient's health status over six months. During the study, socio-demographic data and cost-of-illness data will be recorded. Daxas (tablet) will be administered once daily. The study will provide further data on the safety and tolerability of Daxas.

ELIGIBILITY:
Main Inclusion Criteria:

* severe COPD

Main Exclusion Criteria:

* Child pugh (classified B and C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with severe COPD.
Sampling Method: Non-Probability Sample
Enrollment: 5472 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pre-/post comparison of the COPD status based on patients health status | after 6 months
  Evaluation of treatment success by a COPD-specific patient questionnaire

SECONDARY OUTCOMES:
Effectiveness during treatment | after 6 months
  Evaluation of treatment success by a health status patient questionnaire
Evaluation of tolerability | after 6 months
  assessment of adverse drug reactions
Evaluation of cost-of-illness data | before treatment
  number of consultations, sick leave, hospitalisation, number of and duration of rehab measures
Evaluation of sociodemographic data | before treatment
  employment status, disease management programme
Evaluation of symptom reduction of sputum and cough | after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1699):
- Germany (1699):
  - Nycomed Deutschland GmbH, Aachen
  - Nycomed Deutschland GmbH, Aalen
  - Nycomed Deutschland GmbH, Abensberg
  - Nycomed Deutschland GmbH, Achern
  - Nycomed Deutschland GmbH, Achim
  - Nycomed Deutschland GmbH, Adelebsen
  - Nycomed Deutschland GmbH, Adelsdorf
  - Nycomed Deutschland GmbH, Adenau
  - Nycomed Deutschland GmbH, Adendorf
  - Nycomed Deutschland GmbH, Adorf
  - Nycomed Deutschland GmbH, Ahaus
  - Nycomed Deutschland GmbH, Ahlden
  - Nycomed Deutschland GmbH, Ahlen
  - Nycomed Deutschland GmbH, Ahlerstedt
  - Nycomed Deutschland GmbH, Ahrensburg
  - Nycomed Deutschland GmbH, Ahrensfelde
  - Nycomed Deutschland GmbH, Aichach
  - Nycomed Deutschland GmbH, Aichhalden
  - Nycomed Deutschland GmbH, Aichtal
  - Nycomed Deutschland GmbH, Ainring
  - Nycomed Deutschland GmbH, Aislingen
  - Nycomed Deutschland GmbH, Aken
  - Nycomed Deutschland GmbH, Albstadt
  - Nycomed Deutschland GmbH, Aldenhoven
  - Nycomed Deutschland GmbH, Alfhausen
  - Nycomed Deutschland GmbH, Allersberg
  - Nycomed Deutschland GmbH, Alsbach-Hähnlein
  - Nycomed Deutschland GmbH, Alsdorf
  - Nycomed Deutschland GmbH, Alsenz
  - Nycomed Deutschland GmbH, Altdorf
  - Nycomed Deutschland GmbH, Altena
  - Nycomed Deutschland GmbH, Altenbeken
  - Nycomed Deutschland GmbH, Altenburg
  - Nycomed Deutschland GmbH, Altenholz
  - Nycomed Deutschland GmbH, Altenstadt
  - Nycomed Deutschland GmbH, Altentreptow
  - Nycomed Deutschland GmbH, Althengstett
  - Nycomed Deutschland GmbH, Altlußheim
  - Nycomed Deutschland GmbH, Altötting
  - Nycomed Deutschland GmbH, Altshausen
  - Nycomed Deutschland GmbH, Alzenau in Unterfranken
  - Nycomed Deutschland GmbH, Amberg
  - Nycomed Deutschland GmbH, Amelinghausen
  - Nycomed Deutschland GmbH, Amtsberg
  - Nycomed Deutschland GmbH, Anderbeck
  - Nycomed Deutschland GmbH, Andernach
  - Nycomed Deutschland GmbH, Angersdorf
  - Nycomed Deutschland GmbH, Anhausen
  - Nycomed Deutschland GmbH, Anklam
  - Nycomed Deutschland GmbH, Ankum
  - Nycomed Deutschland GmbH, Annaberg-Buchholz
  - Nycomed Deutschland GmbH, Annweiler am Trifels
  - Nycomed Deutschland GmbH, Ansbach
  - Nycomed Deutschland GmbH, Apen
  - Nycomed Deutschland GmbH, Apolda
  - Nycomed Deutschland GmbH, Appenweier
  - Nycomed Deutschland GmbH, Argenbühl
  - Nycomed Deutschland GmbH, Arneburg
  - Nycomed Deutschland GmbH, Arnsberg
  - Nycomed Deutschland GmbH, Arnschwang
  - Nycomed Deutschland GmbH, Artlenburg
  - Nycomed Deutschland GmbH, Arzberg
  - Nycomed Deutschland GmbH, Asbach
  - Nycomed Deutschland GmbH, Aschaffenburg
  - Nycomed Deutschland GmbH, Aschau A. Inn
  - Nycomed Deutschland GmbH, Aschendorf
  - Nycomed Deutschland GmbH, Aschersleben
  - Nycomed Deutschland GmbH, Aue
  - Nycomed Deutschland GmbH, Auenwald
  - Nycomed Deutschland GmbH, Auerbach
  - Nycomed Deutschland GmbH, Auerbach/Vogtl.
  - Nycomed Deutschland GmbH, Aufkirchen
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Aßlar
  - Nycomed Deutschland GmbH, Babenhausen
  - Nycomed Deutschland GmbH, Babensham
  - Nycomed Deutschland GmbH, Backnang
  - Nycomed Deutschland GmbH, Bad Aibling
  - Nycomed Deutschland GmbH, Bad Bederkesa
  - Nycomed Deutschland GmbH, Bad Belzig
  - Nycomed Deutschland GmbH, Bad Bentheim
  - Nycomed Deutschland GmbH, Bad Berka
  - Nycomed Deutschland GmbH, Bad Bevensen
  - Nycomed Deutschland GmbH, Bad Birnbach
  - Nycomed Deutschland GmbH, Bad Blankenburg
  - Nycomed Deutschland GmbH, Bad Bramstedt
  - Nycomed Deutschland GmbH, Bad Buchau
  - Nycomed Deutschland GmbH, Bad Doberan
  - Nycomed Deutschland GmbH, Bad Driburg
  - Nycomed Deutschland GmbH, Bad Düben
  - Nycomed Deutschland GmbH, Bad Dürrenberg
  - Nycomed Deutschland GmbH, Bad Dürrheim
  - Nycomed Deutschland GmbH, Bad Essen
  - Nycomed Deutschland GmbH, Bad Fallingbostel
  - Nycomed Deutschland GmbH, Bad Feilnbach
  - Nycomed Deutschland GmbH, Bad Freienwalde
  - Nycomed Deutschland GmbH, Bad Friedrichshall
  - Nycomed Deutschland GmbH, Bad Grönenbach
  - Nycomed Deutschland GmbH, Bad Harzburg
  - Nycomed Deutschland GmbH, Bad Homburg
  - Nycomed Deutschland GmbH, Bad Kissingen
  - Nycomed Deutschland GmbH, Bad Klosterlausnitz
  - Nycomed Deutschland GmbH, Bad Kötzting
  - Nycomed Deutschland GmbH, Bad Kreuznach
  - Nycomed Deutschland GmbH, Bad Krozingen
  - Nycomed Deutschland GmbH, Bad Langensalza
  - Nycomed Deutschland GmbH, Bad Lauterberg im Harz
  - Nycomed Deutschland GmbH, Bad Liebenstein
  - Nycomed Deutschland GmbH, Bad Liebenwerda
  - Nycomed Deutschland GmbH, Bad Liebenzell
  - Nycomed Deutschland GmbH, Bad Lippspringe
  - Nycomed Deutschland GmbH, Bad Mergentheim
  - Nycomed Deutschland GmbH, Bad Nauheim
  - Nycomed Deutschland GmbH, Bad Neuenahr-Ahrweiler
  - Nycomed Deutschland GmbH, Bad Neustadt an der Saale
  - Nycomed Deutschland GmbH, Bad Oeynhausen
  - Nycomed Deutschland GmbH, Bad Oldesloe
  - Nycomed Deutschland GmbH, Bad Rappenau
  - Nycomed Deutschland GmbH, Bad Reichenhall
  - Nycomed Deutschland GmbH, Bad Rippoldsau-Schapbach
  - Nycomed Deutschland GmbH, Bad Rothenfelde
  - Nycomed Deutschland GmbH, Bad Saarow
  - Nycomed Deutschland GmbH, Bad Salzuflen
  - Nycomed Deutschland GmbH, Bad Salzungen
  - Nycomed Deutschland GmbH, Bad Schandau
  - Nycomed Deutschland GmbH, Bad Schmiedeberg
  - Nycomed Deutschland GmbH, Bad Schönborn
  - Nycomed Deutschland GmbH, Bad Schussenried
  - Nycomed Deutschland GmbH, Bad Schwalbach
  - Nycomed Deutschland GmbH, Bad Segeberg
  - Nycomed Deutschland GmbH, Bad Staffelstein
  - Nycomed Deutschland GmbH, Bad Sulza
  - Nycomed Deutschland GmbH, Bad Sülze
  - Nycomed Deutschland GmbH, Bad Tennstedt
  - Nycomed Deutschland GmbH, Bad Vilbel
  - Nycomed Deutschland GmbH, Bad Waldsee
  - Nycomed Deutschland GmbH, Bad Wiessee
  - Nycomed Deutschland GmbH, Bad Wildungen
  - Nycomed Deutschland GmbH, Bad Wilsnack
  - Nycomed Deutschland GmbH, Bad Windsheim
  - Nycomed Deutschland GmbH, Bad Wünnenberg
  - Nycomed Deutschland GmbH, Bad Zwischenahn
  - Nycomed Deutschland GmbH, Baden-Baden
  - Nycomed Deutschland GmbH, Badenhausen
  - Nycomed Deutschland GmbH, Baesweiler
  - Nycomed Deutschland GmbH, Bahrdorf
  - Nycomed Deutschland GmbH, Baiersbronn
  - Nycomed Deutschland GmbH, Baindt
  - Nycomed Deutschland GmbH, Bakum
  - Nycomed Deutschland GmbH, Balingen
  - Nycomed Deutschland GmbH, Bamberg
  - Nycomed Deutschland GmbH, Bardowick
  - Nycomed Deutschland GmbH, Bargstedt
  - Nycomed Deutschland GmbH, Barleben
  - Nycomed Deutschland GmbH, Barnstädt
  - Nycomed Deutschland GmbH, Barnstorf
  - Nycomed Deutschland GmbH, Barsinghausen
  - Nycomed Deutschland GmbH, Barth
  - Nycomed Deutschland GmbH, Baruth
  - Nycomed Deutschland GmbH, Barßel
  - Nycomed Deutschland GmbH, Bassenheim
  - Nycomed Deutschland GmbH, Bassum
  - Nycomed Deutschland GmbH, Baunatal
  - Nycomed Deutschland GmbH, Bautzen
  - Nycomed Deutschland GmbH, Bayreuth
  - Nycomed Deutschland GmbH, Beckingen
  - Nycomed Deutschland GmbH, Beckum
  - Nycomed Deutschland GmbH, Beeskow
  - Nycomed Deutschland GmbH, Beilngries
  - Nycomed Deutschland GmbH, Bellheim
  - Nycomed Deutschland GmbH, Belm
  - Nycomed Deutschland GmbH, Bensheim
  - Nycomed Deutschland GmbH, Berching
  - Nycomed Deutschland GmbH, Berchtesgaden
  - Nycomed Deutschland GmbH, Berg
  - Nycomed Deutschland GmbH, Bergen auf Rügen
  - Nycomed Deutschland GmbH, Bergfelde
  - Nycomed Deutschland GmbH, Bergisch Gladbach
  - Nycomed Deutschland GmbH, Bergkamen
  - Nycomed Deutschland GmbH, Bergrheinfeld
  - Nycomed Deutschland GmbH, Bergtheim
  - Nycomed Deutschland GmbH, Berkatal
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Bernau A. Chiemsee
  - Nycomed Deutschland GmbH, Bernburg
  - Nycomed Deutschland GmbH, Bernhardswald
  - Nycomed Deutschland GmbH, Bernkastel-Kues
  - Nycomed Deutschland GmbH, Bernsdorf
  - Nycomed Deutschland GmbH, Bersenbrück
  - Nycomed Deutschland GmbH, Berthelsdorf
  - Nycomed Deutschland GmbH, Beselich
  - Nycomed Deutschland GmbH, Bessenbach
  - Nycomed Deutschland GmbH, Bestensee
  - Nycomed Deutschland GmbH, Bestwig
  - Nycomed Deutschland GmbH, Beucha
  - Nycomed Deutschland GmbH, Bevern
  - Nycomed Deutschland GmbH, Bexbach
  - Nycomed Deutschland GmbH, Biberach
  - Nycomed Deutschland GmbH, Biberach an der Riss
  - Nycomed Deutschland GmbH, Biederitz
  - Nycomed Deutschland GmbH, Bielefeld
  - Nycomed Deutschland GmbH, Bienenbüttel
  - Nycomed Deutschland GmbH, Bietigheim-Bissingen
  - Nycomed Deutschland GmbH, Bingen
  - Nycomed Deutschland GmbH, Bingen am Rhein
  - Nycomed Deutschland GmbH, Binzen
  - Nycomed Deutschland GmbH, Birkenfeld
  - Nycomed Deutschland GmbH, Birkenheide
  - Nycomed Deutschland GmbH, Birresborn
  - Nycomed Deutschland GmbH, Bischofferode
  - Nycomed Deutschland GmbH, Bischofsheim
  - Nycomed Deutschland GmbH, Bischofswerda
  - Nycomed Deutschland GmbH, Bischofswiesen
  - Nycomed Deutschland GmbH, Bismark
  - Nycomed Deutschland GmbH, Bispingen
  - Nycomed Deutschland GmbH, Bitterfeld-Wolfen
  - Nycomed Deutschland GmbH, Blankenhain
  - Nycomed Deutschland GmbH, Blankenrath
  - Nycomed Deutschland GmbH, Blaustein
  - Nycomed Deutschland GmbH, Bleicherode
  - Nycomed Deutschland GmbH, Blumberg
  - Nycomed Deutschland GmbH, Bobritzsch
  - Nycomed Deutschland GmbH, Bocholt
  - Nycomed Deutschland GmbH, Bochum
  - Nycomed Deutschland GmbH, Bodenwöhr
  - Nycomed Deutschland GmbH, Bodman-Ludwigshafen
  - Nycomed Deutschland GmbH, Bogen
  - Nycomed Deutschland GmbH, Bohmte
  - Nycomed Deutschland GmbH, Bonn
  - Nycomed Deutschland GmbH, Bonndorf
  - Nycomed Deutschland GmbH, Boostedt
  - Nycomed Deutschland GmbH, Bopfingen
  - Nycomed Deutschland GmbH, Boppard
  - Nycomed Deutschland GmbH, Borchen
  - Nycomed Deutschland GmbH, Bordesholm
  - Nycomed Deutschland GmbH, Borgentreich
  - Nycomed Deutschland GmbH, Borgholzhausen
  - Nycomed Deutschland GmbH, Borken
  - Nycomed Deutschland GmbH, Borna
  - Nycomed Deutschland GmbH, Bornheim
  - Nycomed Deutschland GmbH, Borsdorf
  - Nycomed Deutschland GmbH, Bous
  - Nycomed Deutschland GmbH, Bovenden
  - Nycomed Deutschland GmbH, Böhlen
  - Nycomed Deutschland GmbH, Bönen
  - Nycomed Deutschland GmbH, Bösingen
  - Nycomed Deutschland GmbH, Bramsche
  - Nycomed Deutschland GmbH, Brand-Erbisdorf
  - Nycomed Deutschland GmbH, Brandenburg
  - Nycomed Deutschland GmbH, Braunschweig
  - Nycomed Deutschland GmbH, Brechen
  - Nycomed Deutschland GmbH, Bredstedt
  - Nycomed Deutschland GmbH, Brehna
  - Nycomed Deutschland GmbH, Breitenbrunn
  - Nycomed Deutschland GmbH, Breitenfelde
  - Nycomed Deutschland GmbH, Bremen
  - Nycomed Deutschland GmbH, Bremerhaven
  - Nycomed Deutschland GmbH, Bretten
  - Nycomed Deutschland GmbH, Brilon
  - Nycomed Deutschland GmbH, Brokstedt
  - Nycomed Deutschland GmbH, Bröckel
  - Nycomed Deutschland GmbH, Bruchköbel
  - Nycomed Deutschland GmbH, Bruchsal
  - Nycomed Deutschland GmbH, Bruck i.d.OPf.
  - Nycomed Deutschland GmbH, Bruckberg
  - Nycomed Deutschland GmbH, Brücken
  - Nycomed Deutschland GmbH, Brühl
  - Nycomed Deutschland GmbH, Buch
  - Nycomed Deutschland GmbH, Buchbach
  - Nycomed Deutschland GmbH, Buckenhof
  - Nycomed Deutschland GmbH, Buckow
  - Nycomed Deutschland GmbH, Burg
  - Nycomed Deutschland GmbH, Burgdorf, Hanover
  - Nycomed Deutschland GmbH, Burgheim
  - Nycomed Deutschland GmbH, Burgstädt
  - Nycomed Deutschland GmbH, Burkhardtsdorf
  - Nycomed Deutschland GmbH, Burow
  - Nycomed Deutschland GmbH, Buttenheim
  - Nycomed Deutschland GmbH, Butzbach
  - Nycomed Deutschland GmbH, Buxheim
  - Nycomed Deutschland GmbH, Büchen
  - Nycomed Deutschland GmbH, Büchenbeuren
  - Nycomed Deutschland GmbH, Bückeburg
  - Nycomed Deutschland GmbH, Büdingen
  - Nycomed Deutschland GmbH, Bühlertann
  - Nycomed Deutschland GmbH, Bünde
  - Nycomed Deutschland GmbH, Büren
  - Nycomed Deutschland GmbH, Bütthard
  - Nycomed Deutschland GmbH, Cadolzburg
  - Nycomed Deutschland GmbH, Calw
  - Nycomed Deutschland GmbH, Castrop-Rauxel
  - Nycomed Deutschland GmbH, Celle
  - Nycomed Deutschland GmbH, Chemnitz
  - Nycomed Deutschland GmbH, Clausthal-Zellerfeld
  - Nycomed Deutschland GmbH, Claußnitz
  - Nycomed Deutschland GmbH, Cloppenburg
  - Nycomed Deutschland GmbH, Coburg
  - Nycomed Deutschland GmbH, Cochem
  - Nycomed Deutschland GmbH, Coesfeld
  - Nycomed Deutschland GmbH, Colditz
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Coswig
  - Nycomed Deutschland GmbH, Cottbus
  - Nycomed Deutschland GmbH, Cölbe
  - Nycomed Deutschland GmbH, Crivitz
  - Nycomed Deutschland GmbH, Cuxhaven
  - Nycomed Deutschland GmbH, Dahlen
  - Nycomed Deutschland GmbH, Dahme
  - Nycomed Deutschland GmbH, Dannstadt-Schauernheim
  - Nycomed Deutschland GmbH, Darmstadt
  - Nycomed Deutschland GmbH, Darscheid
  - Nycomed Deutschland GmbH, Daun
  - Nycomed Deutschland GmbH, Deggendorf
  - Nycomed Deutschland GmbH, Deggingen
  - Nycomed Deutschland GmbH, Delbrück
  - Nycomed Deutschland GmbH, Delitzsch
  - Nycomed Deutschland GmbH, Delmenhorst
  - Nycomed Deutschland GmbH, Demen
  - Nycomed Deutschland GmbH, Demmin
  - Nycomed Deutschland GmbH, Denzlingen
  - Nycomed Deutschland GmbH, Dermbach
  - Nycomed Deutschland GmbH, Dernbach
  - Nycomed Deutschland GmbH, Dessau
  - Nycomed Deutschland GmbH, Detern
  - Nycomed Deutschland GmbH, Detmold
  - Nycomed Deutschland GmbH, Dettenhausen
  - Nycomed Deutschland GmbH, Dettenheim
  - Nycomed Deutschland GmbH, Dettingen an der Erms
  - Nycomed Deutschland GmbH, Dettingen an der Iller
  - Nycomed Deutschland GmbH, Deuben
  - Nycomed Deutschland GmbH, Diedorf
  - Nycomed Deutschland GmbH, Diepenau
  - Nycomed Deutschland GmbH, Diepholz
  - Nycomed Deutschland GmbH, Dietenheim
  - Nycomed Deutschland GmbH, Dietzenbach
  - Nycomed Deutschland GmbH, Dießen am Ammersee
  - Nycomed Deutschland GmbH, Dillingen
  - Nycomed Deutschland GmbH, Dingolfing
  - Nycomed Deutschland GmbH, Dinkelsbühl
  - Nycomed Deutschland GmbH, Dinkelscherben
  - Nycomed Deutschland GmbH, Dinklage
  - Nycomed Deutschland GmbH, Dinslaken
  - Nycomed Deutschland GmbH, Doberlug-Kirchhain
  - Nycomed Deutschland GmbH, Doberschütz
  - Nycomed Deutschland GmbH, Dollern
  - Nycomed Deutschland GmbH, Dommitzsch
  - Nycomed Deutschland GmbH, Donaueschingen
  - Nycomed Deutschland GmbH, Donzdorf
  - Nycomed Deutschland GmbH, Dorfmark
  - Nycomed Deutschland GmbH, Dormagen
  - Nycomed Deutschland GmbH, Dorn-Dürkheim
  - Nycomed Deutschland GmbH, Dornburg
  - Nycomed Deutschland GmbH, Dorndorf-Steudnitz
  - Nycomed Deutschland GmbH, Dorsten
  - Nycomed Deutschland GmbH, Dortmund
  - Nycomed Deutschland GmbH, Dossenheim
  - Nycomed Deutschland GmbH, Döbeln
  - Nycomed Deutschland GmbH, Dörpen
  - Nycomed Deutschland GmbH, Dörzbach
  - Nycomed Deutschland GmbH, Dreetz
  - Nycomed Deutschland GmbH, Drei Gleichen
  - Nycomed Deutschland GmbH, Dreis
  - Nycomed Deutschland GmbH, Dresden
  - Nycomed Deutschland GmbH, Drochtersen
  - Nycomed Deutschland GmbH, Drolshagen
  - Nycomed Deutschland GmbH, Droyßig
  - Nycomed Deutschland GmbH, Dudenhofen
  - Nycomed Deutschland GmbH, Duisburg
  - Nycomed Deutschland GmbH, Dülmen
  - Nycomed Deutschland GmbH, Düren
  - Nycomed Deutschland GmbH, Dürrröhrsdorf
  - Nycomed Deutschland GmbH, Düsseldorf
  - Nycomed Deutschland GmbH, Ebeleben
  - Nycomed Deutschland GmbH, Ebelsbach
  - Nycomed Deutschland GmbH, Ebensfeld
  - Nycomed Deutschland GmbH, Eberbach
  - Nycomed Deutschland GmbH, Ebersdorf B. Coburg
  - Nycomed Deutschland GmbH, Ebrach
  - Nycomed Deutschland GmbH, Eching
  - Nycomed Deutschland GmbH, Eckernförde
  - Nycomed Deutschland GmbH, Edling
  - Nycomed Deutschland GmbH, Effeltrich
  - Nycomed Deutschland GmbH, Egestorf
  - Nycomed Deutschland GmbH, Egg a.d.Günz
  - Nycomed Deutschland GmbH, Eggenstein-Leopoldshafen
  - Nycomed Deutschland GmbH, Eggersdorf
  - Nycomed Deutschland GmbH, Ehingen
  - Nycomed Deutschland GmbH, Ehrenberg
  - Nycomed Deutschland GmbH, Ehringshausen
  - Nycomed Deutschland GmbH, Eichstätt
  - Nycomed Deutschland GmbH, Eicklingen
  - Nycomed Deutschland GmbH, Eilenburg
  - Nycomed Deutschland GmbH, Eimsheim
  - Nycomed Deutschland GmbH, Einbeck
  - Nycomed Deutschland GmbH, Eisenach
  - Nycomed Deutschland GmbH, Eisenhüttenstadt
  - Nycomed Deutschland GmbH, Eisleben Lutherstadt
  - Nycomed Deutschland GmbH, Eitorf
  - Nycomed Deutschland GmbH, Elchesheim
  - Nycomed Deutschland GmbH, Ellefeld
  - Nycomed Deutschland GmbH, Ellerstadt
  - Nycomed Deutschland GmbH, Ellwangen
  - Nycomed Deutschland GmbH, Elmshorn
  - Nycomed Deutschland GmbH, Elsdorf
  - Nycomed Deutschland GmbH, Elsenfeld
  - Nycomed Deutschland GmbH, Elsterwerda
  - Nycomed Deutschland GmbH, Elz
  - Nycomed Deutschland GmbH, Elzach
  - Nycomed Deutschland GmbH, Emden
  - Nycomed Deutschland GmbH, Emleben
  - Nycomed Deutschland GmbH, Emmendingen
  - Nycomed Deutschland GmbH, Emmerich
  - Nycomed Deutschland GmbH, Emmerting
  - Nycomed Deutschland GmbH, Emsdetten
  - Nycomed Deutschland GmbH, Engelskirchen
  - Nycomed Deutschland GmbH, Eningen unter Achalm
  - Nycomed Deutschland GmbH, Enkenbach-Alsenborn
  - Nycomed Deutschland GmbH, Ennepetal
  - Nycomed Deutschland GmbH, Ennigerloh
  - Nycomed Deutschland GmbH, Eppelheim
  - Nycomed Deutschland GmbH, Eppelsheim
  - Nycomed Deutschland GmbH, Eppstein
  - Nycomed Deutschland GmbH, Erding
  - Nycomed Deutschland GmbH, Erftstadt
  - Nycomed Deutschland GmbH, Erfurt
  - Nycomed Deutschland GmbH, Erkelenz
  - Nycomed Deutschland GmbH, Erkner
  - Nycomed Deutschland GmbH, Erlabrunn
  - Nycomed Deutschland GmbH, Erlangen
  - Nycomed Deutschland GmbH, Erlenbach A. Main
  - Nycomed Deutschland GmbH, Erlensee
  - Nycomed Deutschland GmbH, Ermershausen
  - Nycomed Deutschland GmbH, Eschbach
  - Nycomed Deutschland GmbH, Eschelbronn
  - Nycomed Deutschland GmbH, Eschershausen
  - Nycomed Deutschland GmbH, Eschwege
  - Nycomed Deutschland GmbH, Eschweiler
  - Nycomed Deutschland GmbH, Esens
  - Nycomed Deutschland GmbH, Eslohe
  - Nycomed Deutschland GmbH, Espelkamp
  - Nycomed Deutschland GmbH, Espenau
  - Nycomed Deutschland GmbH, Espenhain
  - Nycomed Deutschland GmbH, Essen
  - Nycomed Deutschland GmbH, Essenheim
  - Nycomed Deutschland GmbH, Essingen
  - Nycomed Deutschland GmbH, Ettlingen
  - Nycomed Deutschland GmbH, Euskirchen
  - Nycomed Deutschland GmbH, Falkensee
  - Nycomed Deutschland GmbH, Fellbach
  - Nycomed Deutschland GmbH, Felsberg
  - Nycomed Deutschland GmbH, Feucht
  - Nycomed Deutschland GmbH, Feuchtwangen
  - Nycomed Deutschland GmbH, Filderstadt
  - Nycomed Deutschland GmbH, Finnentrop
  - Nycomed Deutschland GmbH, Finsterwalde
  - Nycomed Deutschland GmbH, Fischbachau
  - Nycomed Deutschland GmbH, Flein
  - Nycomed Deutschland GmbH, Flörsheim-Dalsheim
  - Nycomed Deutschland GmbH, Forbach
  - Nycomed Deutschland GmbH, Forchheim
  - Nycomed Deutschland GmbH, Föhren
  - Nycomed Deutschland GmbH, Framersheim
  - Nycomed Deutschland GmbH, Frankenberg
  - Nycomed Deutschland GmbH, Frankenhardt
  - Nycomed Deutschland GmbH, Frankenthal
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Frankfurt am Main
  - Nycomed Deutschland GmbH, Franzburg
  - Nycomed Deutschland GmbH, Frauenstein
  - Nycomed Deutschland GmbH, Frechen
  - Nycomed Deutschland GmbH, Freiberg
  - Nycomed Deutschland GmbH, Freiburg im Breisgau
  - Nycomed Deutschland GmbH, Freigericht
  - Nycomed Deutschland GmbH, Freilassing
  - Nycomed Deutschland GmbH, Freisen
  - Nycomed Deutschland GmbH, Freital
  - Nycomed Deutschland GmbH, Frensdorf
  - Nycomed Deutschland GmbH, Freudenstadt
  - Nycomed Deutschland GmbH, Freyung
  - Nycomed Deutschland GmbH, Friedberg
  - Nycomed Deutschland GmbH, Friedersdorf
  - Nycomed Deutschland GmbH, Friedland
  - Nycomed Deutschland GmbH, Friedrichshafen
  - Nycomed Deutschland GmbH, Friesack
  - Nycomed Deutschland GmbH, Friesenheim
  - Nycomed Deutschland GmbH, Friesoythe
  - Nycomed Deutschland GmbH, Fröndenberg
  - Nycomed Deutschland GmbH, Fuchsmühl
  - Nycomed Deutschland GmbH, Fulda
  - Nycomed Deutschland GmbH, Fuldatal
  - Nycomed Deutschland GmbH, Furth im Wald
  - Nycomed Deutschland GmbH, Furtwangen im Schwarzwald
  - Nycomed Deutschland GmbH, Fürstenberg
  - Nycomed Deutschland GmbH, Fürstenfeldbruck
  - Nycomed Deutschland GmbH, Fürstenstein
  - Nycomed Deutschland GmbH, Fürstenwalde
  - Nycomed Deutschland GmbH, Fürstenzell
  - Nycomed Deutschland GmbH, Fürth
  - Nycomed Deutschland GmbH, Füssen
  - Nycomed Deutschland GmbH, Gaggenau
  - Nycomed Deutschland GmbH, Gaildorf
  - Nycomed Deutschland GmbH, Gaimersheim
  - Nycomed Deutschland GmbH, Ganderkesee
  - Nycomed Deutschland GmbH, Garbsen
  - Nycomed Deutschland GmbH, Garching a.d.Alz
  - Nycomed Deutschland GmbH, Garmisch-Partenkirchen
  - Nycomed Deutschland GmbH, Garrel
  - Nycomed Deutschland GmbH, Gauting
  - Nycomed Deutschland GmbH, Gebesee
  - Nycomed Deutschland GmbH, Gedern
  - Nycomed Deutschland GmbH, Gefell
  - Nycomed Deutschland GmbH, Gefrees
  - Nycomed Deutschland GmbH, Geisenhausen
  - Nycomed Deutschland GmbH, Geislingen an der Steige
  - Nycomed Deutschland GmbH, Geithain
  - Nycomed Deutschland GmbH, Gelnhausen
  - Nycomed Deutschland GmbH, Gelsenkirchen
  - Nycomed Deutschland GmbH, Gemünden
  - Nycomed Deutschland GmbH, Gensingen
  - Nycomed Deutschland GmbH, Genthin
  - Nycomed Deutschland GmbH, Georgsmarienhütte
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Geretsried
  - Nycomed Deutschland GmbH, Geringswalde
  - Nycomed Deutschland GmbH, Gerlingen
  - Nycomed Deutschland GmbH, Germering
  - Nycomed Deutschland GmbH, Germersheim
  - Nycomed Deutschland GmbH, Gernrode
  - Nycomed Deutschland GmbH, Geroda
  - Nycomed Deutschland GmbH, Gerolstein
  - Nycomed Deutschland GmbH, Gersdorf
  - Nycomed Deutschland GmbH, Gersfeld
  - Nycomed Deutschland GmbH, Gersthofen
  - Nycomed Deutschland GmbH, Geseke
  - Nycomed Deutschland GmbH, Gevelsberg
  - Nycomed Deutschland GmbH, Giessen
  - Nycomed Deutschland GmbH, Gifhorn
  - Nycomed Deutschland GmbH, Gilching
  - Nycomed Deutschland GmbH, Gingen an der Fils
  - Nycomed Deutschland GmbH, Gladbeck
  - Nycomed Deutschland GmbH, Gladenbach
  - Nycomed Deutschland GmbH, Glan-Münchweiler
  - Nycomed Deutschland GmbH, Glauchau
  - Nycomed Deutschland GmbH, Gleichen
  - Nycomed Deutschland GmbH, Glinde
  - Nycomed Deutschland GmbH, Gnoien
  - Nycomed Deutschland GmbH, Gochsheim
  - Nycomed Deutschland GmbH, Goldberg
  - Nycomed Deutschland GmbH, Golzow
  - Nycomed Deutschland GmbH, Gomaringen
  - Nycomed Deutschland GmbH, Gommern
  - Nycomed Deutschland GmbH, Gornau
  - Nycomed Deutschland GmbH, Gornsdorf
  - Nycomed Deutschland GmbH, Goslar
  - Nycomed Deutschland GmbH, Göhren
  - Nycomed Deutschland GmbH, Göllheim
  - Nycomed Deutschland GmbH, Görisried
  - Nycomed Deutschland GmbH, Görlitz
  - Nycomed Deutschland GmbH, Göttingen
  - Nycomed Deutschland GmbH, Grafenau
  - Nycomed Deutschland GmbH, Grafenwöhr
  - Nycomed Deutschland GmbH, Grafing B. München
  - Nycomed Deutschland GmbH, Grafling
  - Nycomed Deutschland GmbH, Gransee
  - Nycomed Deutschland GmbH, Gräfenhainichen
  - Nycomed Deutschland GmbH, Gräfenhausen
  - Nycomed Deutschland GmbH, Gräfenroda
  - Nycomed Deutschland GmbH, Grefrath
  - Nycomed Deutschland GmbH, Greifswald
  - Nycomed Deutschland GmbH, Greiz
  - Nycomed Deutschland GmbH, Greppin
  - Nycomed Deutschland GmbH, Greven
  - Nycomed Deutschland GmbH, Grevenbroich
  - Nycomed Deutschland GmbH, Grimma
  - Nycomed Deutschland GmbH, Gronau
  - Nycomed Deutschland GmbH, Groß Ammensleben
  - Nycomed Deutschland GmbH, Groß Köris
  - Nycomed Deutschland GmbH, Groß Vollstedt
  - Nycomed Deutschland GmbH, Groß Wokern
  - Nycomed Deutschland GmbH, Großbottwar
  - Nycomed Deutschland GmbH, Großen Buseck
  - Nycomed Deutschland GmbH, Großenehrich
  - Nycomed Deutschland GmbH, Großenseebach
  - Nycomed Deutschland GmbH, Großenwiehe
  - Nycomed Deutschland GmbH, Großhansdorf
  - Nycomed Deutschland GmbH, Großheirath
  - Nycomed Deutschland GmbH, Großmaischeid
  - Nycomed Deutschland GmbH, Großröhrsdorf
  - Nycomed Deutschland GmbH, Großschirma
  - Nycomed Deutschland GmbH, Gröbenzell
  - Nycomed Deutschland GmbH, Gröden
  - Nycomed Deutschland GmbH, Grömitz
  - Nycomed Deutschland GmbH, Grub A. Forst
  - Nycomed Deutschland GmbH, Grünbach
  - Nycomed Deutschland GmbH, Grünhainichen
  - Nycomed Deutschland GmbH, Guelders
  - Nycomed Deutschland GmbH, Gummersbach
  - Nycomed Deutschland GmbH, Gundelfingen
  - Nycomed Deutschland GmbH, Gundelsheim
  - Nycomed Deutschland GmbH, Gunzenhausen
  - Nycomed Deutschland GmbH, Gutenberg
  - Nycomed Deutschland GmbH, Güntersleben
  - Nycomed Deutschland GmbH, Güsten
  - Nycomed Deutschland GmbH, Gütersloh
  - Nycomed Deutschland GmbH, Gyhum
  - Nycomed Deutschland GmbH, Haag i.OB
  - Nycomed Deutschland GmbH, Hachenburg
  - Nycomed Deutschland GmbH, Hafenlohr
  - Nycomed Deutschland GmbH, Hagen
  - Nycomed Deutschland GmbH, Hagenow
  - Nycomed Deutschland GmbH, Hainewalde
  - Nycomed Deutschland GmbH, Haiterbach
  - Nycomed Deutschland GmbH, Halbendorf
  - Nycomed Deutschland GmbH, Haldensleben I
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Halsbrücke
  - Nycomed Deutschland GmbH, Haltern am See
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Hamelin
  - Nycomed Deutschland GmbH, Hamm
  - Nycomed Deutschland GmbH, Hammelburg
  - Nycomed Deutschland GmbH, Hamminkeln
  - Nycomed Deutschland GmbH, Hanau
  - Nycomed Deutschland GmbH, Hanover
  - Nycomed Deutschland GmbH, Hardheim
  - Nycomed Deutschland GmbH, Harsewinkel
  - Nycomed Deutschland GmbH, Hartenstein
  - Nycomed Deutschland GmbH, Harthausen
  - Nycomed Deutschland GmbH, Haslach im Kinzigtal
  - Nycomed Deutschland GmbH, Hattingen
  - Nycomed Deutschland GmbH, Haunsheim
  - Nycomed Deutschland GmbH, Hausham
  - Nycomed Deutschland GmbH, Hauzenberg
  - Nycomed Deutschland GmbH, Haßloch
  - Nycomed Deutschland GmbH, Haßmersheim
  - Nycomed Deutschland GmbH, Heckelberg-Brunow
  - Nycomed Deutschland GmbH, Hecklingen
  - Nycomed Deutschland GmbH, Heddesheim
  - Nycomed Deutschland GmbH, Hedersleben
  - Nycomed Deutschland GmbH, Heek
  - Nycomed Deutschland GmbH, Heiddorf
  - Nycomed Deutschland GmbH, Heideck
  - Nycomed Deutschland GmbH, Heidelberg
  - Nycomed Deutschland GmbH, Heidenheim
  - Nycomed Deutschland GmbH, Heilbronn
  - Nycomed Deutschland GmbH, Heiligenhaus
  - Nycomed Deutschland GmbH, Heilsbronn
  - Nycomed Deutschland GmbH, Heinsberg
  - Nycomed Deutschland GmbH, Hellenthal
  - Nycomed Deutschland GmbH, Helmbrechts
  - Nycomed Deutschland GmbH, Helmstedt
  - Nycomed Deutschland GmbH, Hemau
  - Nycomed Deutschland GmbH, Hemer
  - Nycomed Deutschland GmbH, Hemmersheim
  - Nycomed Deutschland GmbH, Hemmoor
  - Nycomed Deutschland GmbH, Hemsbach
  - Nycomed Deutschland GmbH, Henstedt-Ulzburg
  - Nycomed Deutschland GmbH, Herbolzheim
  - Nycomed Deutschland GmbH, Herborn
  - Nycomed Deutschland GmbH, Herbrechtingen
  - Nycomed Deutschland GmbH, Herbstein
  - Nycomed Deutschland GmbH, Hermsdorf
  - Nycomed Deutschland GmbH, Herne
  - Nycomed Deutschland GmbH, Heroldsberg
  - Nycomed Deutschland GmbH, Herrenberg
  - Nycomed Deutschland GmbH, Herscheid
  - Nycomed Deutschland GmbH, Herten
  - Nycomed Deutschland GmbH, Herzberg
  - Nycomed Deutschland GmbH, Herzberg am Harz
  - Nycomed Deutschland GmbH, Herzogenaurach
  - Nycomed Deutschland GmbH, Herzogenrath
  - Nycomed Deutschland GmbH, Heuchlingen
  - Nycomed Deutschland GmbH, Heyerode
  - Nycomed Deutschland GmbH, Heßdorf
  - Nycomed Deutschland GmbH, Hildesheim
  - Nycomed Deutschland GmbH, Hille
  - Nycomed Deutschland GmbH, Hilpoltstein
  - Nycomed Deutschland GmbH, Hilzingen
  - Nycomed Deutschland GmbH, Hinterhermsdorf
  - Nycomed Deutschland GmbH, Hirschau
  - Nycomed Deutschland GmbH, Hirschberg an der Bergstraße
  - Nycomed Deutschland GmbH, Hirschstein
  - Nycomed Deutschland GmbH, Hitzacker
  - Nycomed Deutschland GmbH, Hochheim am Main
  - Nycomed Deutschland GmbH, Hof
  - Nycomed Deutschland GmbH, Hofbieber
  - Nycomed Deutschland GmbH, Hofheim am Taunus
  - Nycomed Deutschland GmbH, Hohberg
  - Nycomed Deutschland GmbH, Hohen Neuendorf
  - Nycomed Deutschland GmbH, Hohenbocka
  - Nycomed Deutschland GmbH, Hohenbrunn
  - Nycomed Deutschland GmbH, Hohenfels
  - Nycomed Deutschland GmbH, Hohenpeißenberg
  - Nycomed Deutschland GmbH, Hoisdorf
  - Nycomed Deutschland GmbH, Holzdorf
  - Nycomed Deutschland GmbH, Holzheim
  - Nycomed Deutschland GmbH, Holzkirchen
  - Nycomed Deutschland GmbH, Holzweißig
  - Nycomed Deutschland GmbH, Homburg
  - Nycomed Deutschland GmbH, Hoppegarten
  - Nycomed Deutschland GmbH, Hopsten
  - Nycomed Deutschland GmbH, Hornburg
  - Nycomed Deutschland GmbH, Horstmar
  - Nycomed Deutschland GmbH, Hosena
  - Nycomed Deutschland GmbH, Hoyerswerda
  - Nycomed Deutschland GmbH, Höchenschwand
  - Nycomed Deutschland GmbH, Höchstadt a.d.Aisch
  - Nycomed Deutschland GmbH, Höhn
  - Nycomed Deutschland GmbH, Höhr-Grenzhausen
  - Nycomed Deutschland GmbH, Hörstel
  - Nycomed Deutschland GmbH, Hövelhof
  - Nycomed Deutschland GmbH, Höxter
  - Nycomed Deutschland GmbH, Hude
  - Nycomed Deutschland GmbH, Huglfing
  - Nycomed Deutschland GmbH, Hummeltal
  - Nycomed Deutschland GmbH, Huska
  - Nycomed Deutschland GmbH, Hückelhoven
  - Nycomed Deutschland GmbH, Hückeswagen
  - Nycomed Deutschland GmbH, Hüffenhardt
  - Nycomed Deutschland GmbH, Hüllhorst
  - Nycomed Deutschland GmbH, Hünfeld
  - Nycomed Deutschland GmbH, Hünfelden
  - Nycomed Deutschland GmbH, Hürth
  - Nycomed Deutschland GmbH, Ibbenbueren
  - Nycomed Deutschland GmbH, Ichtershausen
  - Nycomed Deutschland GmbH, Idar-Oberstein
  - Nycomed Deutschland GmbH, Ifta
  - Nycomed Deutschland GmbH, Igensdorf
  - Nycomed Deutschland GmbH, Ilmenau
  - Nycomed Deutschland GmbH, Ilvesheim
  - Nycomed Deutschland GmbH, Ingolstadt
  - Nycomed Deutschland GmbH, Inning A. Ammersee
  - Nycomed Deutschland GmbH, Inning A. Holz
  - Nycomed Deutschland GmbH, Iserlohn
  - Nycomed Deutschland GmbH, Ismaning
  - Nycomed Deutschland GmbH, Isselburg
  - Nycomed Deutschland GmbH, Issum
  - Nycomed Deutschland GmbH, Itzehoe
  - Nycomed Deutschland GmbH, Jena
  - Nycomed Deutschland GmbH, Jerichow
  - Nycomed Deutschland GmbH, Jessen
  - Nycomed Deutschland GmbH, Jever
  - Nycomed Deutschland GmbH, Jüchen
  - Nycomed Deutschland GmbH, Jüterbog
  - Nycomed Deutschland GmbH, Kahl A. Main
  - Nycomed Deutschland GmbH, Kaiserslautern
  - Nycomed Deutschland GmbH, Kamen
  - Nycomed Deutschland GmbH, Kamenz
  - Nycomed Deutschland GmbH, Kapellendorf
  - Nycomed Deutschland GmbH, Karben
  - Nycomed Deutschland GmbH, Karlsfeld
  - Nycomed Deutschland GmbH, Karlsruhe
  - Nycomed Deutschland GmbH, Kassel
  - Nycomed Deutschland GmbH, Kastl
  - Nycomed Deutschland GmbH, Katzhütte
  - Nycomed Deutschland GmbH, Kaufbeuren
  - Nycomed Deutschland GmbH, Kaulsdorf
  - Nycomed Deutschland GmbH, Kämpfelbach
  - Nycomed Deutschland GmbH, Kehl
  - Nycomed Deutschland GmbH, Kelheim
  - Nycomed Deutschland GmbH, Kelkheim
  - Nycomed Deutschland GmbH, Kemberg
  - Nycomed Deutschland GmbH, Kemnitz
  - Nycomed Deutschland GmbH, Kempen
  - Nycomed Deutschland GmbH, Kempenich
  - Nycomed Deutschland GmbH, Kempfeld
  - Nycomed Deutschland GmbH, Kempten
  - Nycomed Deutschland GmbH, Kenzingen
  - Nycomed Deutschland GmbH, Kerken
  - Nycomed Deutschland GmbH, Kernen Im Remstal
  - Nycomed Deutschland GmbH, Kiel
  - Nycomed Deutschland GmbH, Kierspe
  - Nycomed Deutschland GmbH, Kindsbach
  - Nycomed Deutschland GmbH, Kippenheim
  - Nycomed Deutschland GmbH, Kirchberg
  - Nycomed Deutschland GmbH, Kirchhain
  - Nycomed Deutschland GmbH, Kirchham
  - Nycomed Deutschland GmbH, Kirchheilingen
  - Nycomed Deutschland GmbH, Kirchheim B. München
  - Nycomed Deutschland GmbH, Kirchhundem
  - Nycomed Deutschland GmbH, Kirchlengern
  - Nycomed Deutschland GmbH, Kirn
  - Nycomed Deutschland GmbH, Kisselbach
  - Nycomed Deutschland GmbH, Kißlegg
  - Nycomed Deutschland GmbH, Kleines Wiesental
  - Nycomed Deutschland GmbH, Kleinheubach
  - Nycomed Deutschland GmbH, Kleinwallstadt
  - Nycomed Deutschland GmbH, Kleve
  - Nycomed Deutschland GmbH, Klingenthal
  - Nycomed Deutschland GmbH, Knittlingen
  - Nycomed Deutschland GmbH, Koblenz
  - Nycomed Deutschland GmbH, Kolbermoor
  - Nycomed Deutschland GmbH, Konstanz
  - Nycomed Deutschland GmbH, Konzell
  - Nycomed Deutschland GmbH, Korschenbroich
  - Nycomed Deutschland GmbH, Königs Wusterhausen
  - Nycomed Deutschland GmbH, Königsbrunn
  - Nycomed Deutschland GmbH, Königsbrück
  - Nycomed Deutschland GmbH, Königsee
  - Nycomed Deutschland GmbH, Königstein im Taunus
  - Nycomed Deutschland GmbH, Königstein/Sächs. Schw.
  - Nycomed Deutschland GmbH, Königswinter
  - Nycomed Deutschland GmbH, Köthen
  - Nycomed Deutschland GmbH, Kraiburg A. Inn
  - Nycomed Deutschland GmbH, Krefeld
  - Nycomed Deutschland GmbH, Kremmen
  - Nycomed Deutschland GmbH, Kressbronn am Bodensee
  - Nycomed Deutschland GmbH, Kreuztal
  - Nycomed Deutschland GmbH, Kronberg
  - Nycomed Deutschland GmbH, Kronshagen
  - Nycomed Deutschland GmbH, Krumpa
  - Nycomed Deutschland GmbH, Kuchen
  - Nycomed Deutschland GmbH, Kuhardt
  - Nycomed Deutschland GmbH, Kulmbach
  - Nycomed Deutschland GmbH, Kurort Seiffen
  - Nycomed Deutschland GmbH, Kusel
  - Nycomed Deutschland GmbH, Kühbach
  - Nycomed Deutschland GmbH, Künzelsau
  - Nycomed Deutschland GmbH, Kürnbach
  - Nycomed Deutschland GmbH, Kyllburg
  - Nycomed Deutschland GmbH, Kyritz
  - Nycomed Deutschland GmbH, Ladbergen
  - Nycomed Deutschland GmbH, Lahnau
  - Nycomed Deutschland GmbH, Laichingen
  - Nycomed Deutschland GmbH, Lalling
  - Nycomed Deutschland GmbH, Lamstedt
  - Nycomed Deutschland GmbH, Landau
  - Nycomed Deutschland GmbH, Landau a.d.Isar
  - Nycomed Deutschland GmbH, Landesbergen
  - Nycomed Deutschland GmbH, Landsberg
  - Nycomed Deutschland GmbH, Landsberg am Lech
  - Nycomed Deutschland GmbH, Landshut
  - Nycomed Deutschland GmbH, Langen
  - Nycomed Deutschland GmbH, Langenargen
  - Nycomed Deutschland GmbH, Langenberg
  - Nycomed Deutschland GmbH, Langenbrettach
  - Nycomed Deutschland GmbH, Langendorf
  - Nycomed Deutschland GmbH, Langenfeld
  - Nycomed Deutschland GmbH, Langenleuba-Niederhain
  - Nycomed Deutschland GmbH, Langerwehe
  - Nycomed Deutschland GmbH, Langula
  - Nycomed Deutschland GmbH, Langweid A. Lech
  - Nycomed Deutschland GmbH, Lauchhammer
  - Nycomed Deutschland GmbH, Lauchringen
  - Nycomed Deutschland GmbH, Lauenburg
  - Nycomed Deutschland GmbH, Laufen
  - Nycomed Deutschland GmbH, Lauingen
  - Nycomed Deutschland GmbH, Lauter
  - Nycomed Deutschland GmbH, Lauterbach
  - Nycomed Deutschland GmbH, Lautertal
  - Nycomed Deutschland GmbH, Lähden
  - Nycomed Deutschland GmbH, Lebach
  - Nycomed Deutschland GmbH, Lebus
  - Nycomed Deutschland GmbH, Leer
  - Nycomed Deutschland GmbH, Legefeld
  - Nycomed Deutschland GmbH, Leimersheim
  - Nycomed Deutschland GmbH, Leinburg
  - Nycomed Deutschland GmbH, Leipheim
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Leisnig
  - Nycomed Deutschland GmbH, Lemberg
  - Nycomed Deutschland GmbH, Lemförde
  - Nycomed Deutschland GmbH, Lennestadt
  - Nycomed Deutschland GmbH, Lensahn
  - Nycomed Deutschland GmbH, Leonberg
  - Nycomed Deutschland GmbH, Letschin
  - Nycomed Deutschland GmbH, Leuna
  - Nycomed Deutschland GmbH, Leutenbach
  - Nycomed Deutschland GmbH, Leutershausen
  - Nycomed Deutschland GmbH, Leverkusen
  - Nycomed Deutschland GmbH, Lichtenberg
  - Nycomed Deutschland GmbH, Lichtenfels
  - Nycomed Deutschland GmbH, Lienen
  - Nycomed Deutschland GmbH, Limbach-Oberfrohna
  - Nycomed Deutschland GmbH, Limburgerhof
  - Nycomed Deutschland GmbH, Linden
  - Nycomed Deutschland GmbH, Lindenfels
  - Nycomed Deutschland GmbH, Lindow
  - Nycomed Deutschland GmbH, Lingenfeld
  - Nycomed Deutschland GmbH, Lippetal
  - Nycomed Deutschland GmbH, Lippstadt
  - Nycomed Deutschland GmbH, Lisberg
  - Nycomed Deutschland GmbH, Litzendorf
  - Nycomed Deutschland GmbH, Lobstädt
  - Nycomed Deutschland GmbH, Lohmar
  - Nycomed Deutschland GmbH, Lohr a. Main
  - Nycomed Deutschland GmbH, Lohra
  - Nycomed Deutschland GmbH, Lohsa
  - Nycomed Deutschland GmbH, Lollar
  - Nycomed Deutschland GmbH, Lonsee
  - Nycomed Deutschland GmbH, Lorch
  - Nycomed Deutschland GmbH, Losheim
  - Nycomed Deutschland GmbH, Loxstedt
  - Nycomed Deutschland GmbH, Loßburg
  - Nycomed Deutschland GmbH, Löbejün
  - Nycomed Deutschland GmbH, Löffingen
  - Nycomed Deutschland GmbH, Löhne
  - Nycomed Deutschland GmbH, Lubmin
  - Nycomed Deutschland GmbH, Luckenwalde
  - Nycomed Deutschland GmbH, Ludwigsburg
  - Nycomed Deutschland GmbH, Ludwigshafen am Rhein
  - Nycomed Deutschland GmbH, Ludwigsstadt
  - Nycomed Deutschland GmbH, Lübbecke
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Lüdenscheid
  - Nycomed Deutschland GmbH, Lügde
  - Nycomed Deutschland GmbH, Lüneburg
  - Nycomed Deutschland GmbH, Lünen
  - Nycomed Deutschland GmbH, Lüssow
  - Nycomed Deutschland GmbH, Lützow
  - Nycomed Deutschland GmbH, Lychen
  - Nycomed Deutschland GmbH, Machern
  - Nycomed Deutschland GmbH, Magdeburg
  - Nycomed Deutschland GmbH, Magstadt
  - Nycomed Deutschland GmbH, Maikammer
  - Nycomed Deutschland GmbH, Mainaschaff
  - Nycomed Deutschland GmbH, Mainleus
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Malchin
  - Nycomed Deutschland GmbH, Malsch
  - Nycomed Deutschland GmbH, Mamming
  - Nycomed Deutschland GmbH, Mandelbachtal
  - Nycomed Deutschland GmbH, Mannheim
  - Nycomed Deutschland GmbH, Marbach am Neckar
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Marienberg
  - Nycomed Deutschland GmbH, Markdorf
  - Nycomed Deutschland GmbH, Markersdorf
  - Nycomed Deutschland GmbH, Markkleeberg
  - Nycomed Deutschland GmbH, Marklohe
  - Nycomed Deutschland GmbH, Markranstädt
  - Nycomed Deutschland GmbH, Markt Bibart
  - Nycomed Deutschland GmbH, Markt Schwaben
  - Nycomed Deutschland GmbH, Marktheidenfeld
  - Nycomed Deutschland GmbH, Marktl
  - Nycomed Deutschland GmbH, Marktleugast
  - Nycomed Deutschland GmbH, Marktoberdorf
  - Nycomed Deutschland GmbH, Marl
  - Nycomed Deutschland GmbH, Marne
  - Nycomed Deutschland GmbH, Marnitz
  - Nycomed Deutschland GmbH, Maulburg
  - Nycomed Deutschland GmbH, Maxdorf
  - Nycomed Deutschland GmbH, Mayen
  - Nycomed Deutschland GmbH, Maßweiler
  - Nycomed Deutschland GmbH, Märkisch Buchholz
  - Nycomed Deutschland GmbH, Märkische Heide
  - Nycomed Deutschland GmbH, Meckenheim
  - Nycomed Deutschland GmbH, Medebach
  - Nycomed Deutschland GmbH, Meeder
  - Nycomed Deutschland GmbH, Meerane
  - Nycomed Deutschland GmbH, Meerbusch
  - Nycomed Deutschland GmbH, Mehren
  - Nycomed Deutschland GmbH, Mehrstetten
  - Nycomed Deutschland GmbH, Meine
  - Nycomed Deutschland GmbH, Meinersen
  - Nycomed Deutschland GmbH, Meitingen
  - Nycomed Deutschland GmbH, Meißen
  - Nycomed Deutschland GmbH, Meißenheim
  - Nycomed Deutschland GmbH, Melle
  - Nycomed Deutschland GmbH, Melsungen
  - Nycomed Deutschland GmbH, Memmelsdorf
  - Nycomed Deutschland GmbH, Menden
  - Nycomed Deutschland GmbH, Mendig
  - Nycomed Deutschland GmbH, Mengen
  - Nycomed Deutschland GmbH, Mengersgereuth-Hämmern
  - Nycomed Deutschland GmbH, Merchweiler
  - Nycomed Deutschland GmbH, Merkendorf
  - Nycomed Deutschland GmbH, Merseburg
  - Nycomed Deutschland GmbH, Merxheim
  - Nycomed Deutschland GmbH, Merzenich
  - Nycomed Deutschland GmbH, Merzig
  - Nycomed Deutschland GmbH, Messkirch
  - Nycomed Deutschland GmbH, Metelen
  - Nycomed Deutschland GmbH, Mettlach
  - Nycomed Deutschland GmbH, Miesbach
  - Nycomed Deutschland GmbH, Mihla
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, Mirow
  - Nycomed Deutschland GmbH, Mittelbach
  - Nycomed Deutschland GmbH, Mittenwald
  - Nycomed Deutschland GmbH, Mittweida
  - Nycomed Deutschland GmbH, Moers
  - Nycomed Deutschland GmbH, Molfsee
  - Nycomed Deutschland GmbH, Monheim
  - Nycomed Deutschland GmbH, Monheim am Rhein
  - Nycomed Deutschland GmbH, Monschau
  - Nycomed Deutschland GmbH, Montabaur
  - Nycomed Deutschland GmbH, Moosinning
  - Nycomed Deutschland GmbH, Morbach
  - Nycomed Deutschland GmbH, Mosbach
  - Nycomed Deutschland GmbH, Möckmühl
  - Nycomed Deutschland GmbH, Möhnesee
  - Nycomed Deutschland GmbH, Mölln
  - Nycomed Deutschland GmbH, Mömbris
  - Nycomed Deutschland GmbH, Mönchengladbach
  - Nycomed Deutschland GmbH, Mönchsroth
  - Nycomed Deutschland GmbH, Mönchweiler
  - Nycomed Deutschland GmbH, Mörfelden-Walldorf
  - Nycomed Deutschland GmbH, Mudersbach
  - Nycomed Deutschland GmbH, Mutzschen
  - Nycomed Deutschland GmbH, Mücheln
  - Nycomed Deutschland GmbH, Mühlacker
  - Nycomed Deutschland GmbH, Mühlau
  - Nycomed Deutschland GmbH, Mühldorf A. Inn
  - Nycomed Deutschland GmbH, Mühlhausen
  - Nycomed Deutschland GmbH, Mühltroff
  - Nycomed Deutschland GmbH, Mülheim
  - Nycomed Deutschland GmbH, Mülsen
  - Nycomed Deutschland GmbH, Münchberg
  - Nycomed Deutschland GmbH, Müncheberg
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münchweiler an der Rodalb
  - Nycomed Deutschland GmbH, Münster
  - Nycomed Deutschland GmbH, Mylau
  - Nycomed Deutschland GmbH, Nabburg
  - Nycomed Deutschland GmbH, Nackenheim
  - Nycomed Deutschland GmbH, Nagold
  - Nycomed Deutschland GmbH, Nalbach
  - Nycomed Deutschland GmbH, Nastätten
  - Nycomed Deutschland GmbH, Naumburg
  - Nycomed Deutschland GmbH, Naunhof
  - Nycomed Deutschland GmbH, Neckargemünd
  - Nycomed Deutschland GmbH, Neetze
  - Nycomed Deutschland GmbH, Netphen
  - Nycomed Deutschland GmbH, Nettetal
  - Nycomed Deutschland GmbH, Neu-Ulm
  - Nycomed Deutschland GmbH, Neubiberg
  - Nycomed Deutschland GmbH, Neubrandenburg
  - Nycomed Deutschland GmbH, Neuburg a.Inn
  - Nycomed Deutschland GmbH, Neuburg an der Donau
  - Nycomed Deutschland GmbH, Neuenburg am Rhein
  - Nycomed Deutschland GmbH, Neuenhagen
  - Nycomed Deutschland GmbH, Neuenkirchen-Vörden
  - Nycomed Deutschland GmbH, Neuenrade
  - Nycomed Deutschland GmbH, Neugersdorf
  - Nycomed Deutschland GmbH, Neuhausen ob Eck
  - Nycomed Deutschland GmbH, Neukirch/Lausitz
  - Nycomed Deutschland GmbH, Neukirchen beim Heiligen Blut
  - Nycomed Deutschland GmbH, Neukirchen-Vluyn
  - Nycomed Deutschland GmbH, Neuler
  - Nycomed Deutschland GmbH, Neumünster
  - Nycomed Deutschland GmbH, Neunburg vorm Wald
  - Nycomed Deutschland GmbH, Neunkirchen
  - Nycomed Deutschland GmbH, Neuötting
  - Nycomed Deutschland GmbH, Neuried
  - Nycomed Deutschland GmbH, Neuruppin
  - Nycomed Deutschland GmbH, Neusorg
  - Nycomed Deutschland GmbH, Neuss
  - Nycomed Deutschland GmbH, Neustadt
  - Nycomed Deutschland GmbH, Neustadt a.d.Aisch
  - Nycomed Deutschland GmbH, Neustadt an der Donau
  - Nycomed Deutschland GmbH, Neustadt an der Orla
  - Nycomed Deutschland GmbH, Neustadt an der Weinstraße
  - Nycomed Deutschland GmbH, Neustadt B. Coburg
  - Nycomed Deutschland GmbH, Neustadt in Sachsen
  - Nycomed Deutschland GmbH, Neustadt-Glewe
  - Nycomed Deutschland GmbH, Neustadt/Harz
  - Nycomed Deutschland GmbH, Neuwied
  - Nycomed Deutschland GmbH, Newel
  - Nycomed Deutschland GmbH, Nidda
  - Nycomed Deutschland GmbH, Nidderau
  - Nycomed Deutschland GmbH, Nieder-Olm
  - Nycomed Deutschland GmbH, Niederdorla
  - Nycomed Deutschland GmbH, Niederkassel
  - Nycomed Deutschland GmbH, Niepars
  - Nycomed Deutschland GmbH, Niestetal
  - Nycomed Deutschland GmbH, Nobitz
  - Nycomed Deutschland GmbH, Nohfelden
  - Nycomed Deutschland GmbH, Norderstedt
  - Nycomed Deutschland GmbH, Nordheim
  - Nycomed Deutschland GmbH, Nordholz
  - Nycomed Deutschland GmbH, Nordhorn
  - Nycomed Deutschland GmbH, Nordstrand
  - Nycomed Deutschland GmbH, Nortorf
  - Nycomed Deutschland GmbH, Nossen
  - Nycomed Deutschland GmbH, Nördlingen
  - Nycomed Deutschland GmbH, Nörten-Hardenberg
  - Nycomed Deutschland GmbH, Nuremberg
  - Nycomed Deutschland GmbH, Nußloch
  - Nycomed Deutschland GmbH, Ober-Ramstadt
  - Nycomed Deutschland GmbH, Oberaudorf
  - Nycomed Deutschland GmbH, Obercunnersdorf
  - Nycomed Deutschland GmbH, Oberdorla
  - Nycomed Deutschland GmbH, Obergurig
  - Nycomed Deutschland GmbH, Oberhaching
  - Nycomed Deutschland GmbH, Oberhausen
  - Nycomed Deutschland GmbH, Oberkirch
  - Nycomed Deutschland GmbH, Oberkochen
  - Nycomed Deutschland GmbH, Oberkrämer
  - Nycomed Deutschland GmbH, Obermichelbach
  - Nycomed Deutschland GmbH, Oberndorf Am Neckar
  - Nycomed Deutschland GmbH, Obernzenn
  - Nycomed Deutschland GmbH, Oberried
  - Nycomed Deutschland GmbH, Obertshausen
  - Nycomed Deutschland GmbH, Oberursel
  - Nycomed Deutschland GmbH, Ochtendung
  - Nycomed Deutschland GmbH, Ochtrup
  - Nycomed Deutschland GmbH, Odenthal
  - Nycomed Deutschland GmbH, Oderwitz
  - Nycomed Deutschland GmbH, Oederan
  - Nycomed Deutschland GmbH, Oelde
  - Nycomed Deutschland GmbH, Oer-Erkenschwick
  - Nycomed Deutschland GmbH, Oerel
  - Nycomed Deutschland GmbH, Oerlinghausen
  - Nycomed Deutschland GmbH, Oettingen i.Bay.
  - Nycomed Deutschland GmbH, Offenbach
  - Nycomed Deutschland GmbH, Offenbach an der Queich
  - Nycomed Deutschland GmbH, Offenburg
  - Nycomed Deutschland GmbH, Oftersheim
  - Nycomed Deutschland GmbH, Olbernhau
  - Nycomed Deutschland GmbH, Olbersdorf
  - Nycomed Deutschland GmbH, Olching
  - Nycomed Deutschland GmbH, Oldenburg
  - Nycomed Deutschland GmbH, Oldenburg in Holstein
  - Nycomed Deutschland GmbH, Oldenswort
  - Nycomed Deutschland GmbH, Olfen
  - Nycomed Deutschland GmbH, Olpe
  - Nycomed Deutschland GmbH, Oranienbaum
  - Nycomed Deutschland GmbH, Oranienburg
  - Nycomed Deutschland GmbH, Ortenberg
  - Nycomed Deutschland GmbH, Oschatz
  - Nycomed Deutschland GmbH, Osnabrück
  - Nycomed Deutschland GmbH, Osten
  - Nycomed Deutschland GmbH, Osterburg
  - Nycomed Deutschland GmbH, Osterhofen
  - Nycomed Deutschland GmbH, Osternienburg
  - Nycomed Deutschland GmbH, Ostfildern
  - Nycomed Deutschland GmbH, Osthofen
  - Nycomed Deutschland GmbH, Ostrach
  - Nycomed Deutschland GmbH, Ostrhauderfehn
  - Nycomed Deutschland GmbH, Ostseebad Binz
  - Nycomed Deutschland GmbH, Ostseebad Boltenhagen
  - Nycomed Deutschland GmbH, Ottendorf
  - Nycomed Deutschland GmbH, Ottendorf-Okrilla
  - Nycomed Deutschland GmbH, Otterbach
  - Nycomed Deutschland GmbH, Otterndorf
  - Nycomed Deutschland GmbH, Ottobeuren
  - Nycomed Deutschland GmbH, Ottobrunn bei München
  - Nycomed Deutschland GmbH, Overath
  - Nycomed Deutschland GmbH, Oy-Mittelberg
  - Nycomed Deutschland GmbH, Öhningen
  - Nycomed Deutschland GmbH, Östringen
  - Nycomed Deutschland GmbH, Paderborn
  - Nycomed Deutschland GmbH, Panschwitz-Kuckau
  - Nycomed Deutschland GmbH, Papenburg
  - Nycomed Deutschland GmbH, Parsberg
  - Nycomed Deutschland GmbH, Passau
  - Nycomed Deutschland GmbH, Peiting
  - Nycomed Deutschland GmbH, Penig
  - Nycomed Deutschland GmbH, Penzberg
  - Nycomed Deutschland GmbH, Perleberg
  - Nycomed Deutschland GmbH, Petershagen
  - Nycomed Deutschland GmbH, Pfakofen
  - Nycomed Deutschland GmbH, Pforzheim
  - Nycomed Deutschland GmbH, Pfullendorf
  - Nycomed Deutschland GmbH, Pfullingen
  - Nycomed Deutschland GmbH, Philippsburg
  - Nycomed Deutschland GmbH, Pilsting
  - Nycomed Deutschland GmbH, Pinneberg
  - Nycomed Deutschland GmbH, Pirmasens
  - Nycomed Deutschland GmbH, Pirna
  - Nycomed Deutschland GmbH, Plankstadt
  - Nycomed Deutschland GmbH, Plau am See
  - Nycomed Deutschland GmbH, Plauen
  - Nycomed Deutschland GmbH, Pleidelsheim
  - Nycomed Deutschland GmbH, Pleiskirchen
  - Nycomed Deutschland GmbH, Plettenberg
  - Nycomed Deutschland GmbH, Pleystein
  - Nycomed Deutschland GmbH, Plön
  - Nycomed Deutschland GmbH, Plüderhausen
  - Nycomed Deutschland GmbH, Pockau
  - Nycomed Deutschland GmbH, Poing
  - Nycomed Deutschland GmbH, Polch
  - Nycomed Deutschland GmbH, Poppenhausen
  - Nycomed Deutschland GmbH, Porta Westfalica
  - Nycomed Deutschland GmbH, Potsdam
  - Nycomed Deutschland GmbH, Pöttmes
  - Nycomed Deutschland GmbH, Pößneck
  - Nycomed Deutschland GmbH, Preetz
  - Nycomed Deutschland GmbH, Premnitz
  - Nycomed Deutschland GmbH, Pretzfeld
  - Nycomed Deutschland GmbH, Preußisch Oldendorf
  - Nycomed Deutschland GmbH, Priestewitz
  - Nycomed Deutschland GmbH, Pulheim
  - Nycomed Deutschland GmbH, Pullach I. Isartal
  - Nycomed Deutschland GmbH, Pulsnitz
  - Nycomed Deutschland GmbH, Putbus
  - Nycomed Deutschland GmbH, Quakenbrück
  - Nycomed Deutschland GmbH, Queidersbach
  - Nycomed Deutschland GmbH, Radeberg
  - Nycomed Deutschland GmbH, Radebeul
  - Nycomed Deutschland GmbH, Radeburg
  - Nycomed Deutschland GmbH, Radevormwald
  - Nycomed Deutschland GmbH, Radolfzell
  - Nycomed Deutschland GmbH, Raguhn
  - Nycomed Deutschland GmbH, Rahden
  - Nycomed Deutschland GmbH, Rain
  - Nycomed Deutschland GmbH, Ralbitz-Rosenthal
  - Nycomed Deutschland GmbH, Ramsen
  - Nycomed Deutschland GmbH, Ramstein-Miesenbach
  - Nycomed Deutschland GmbH, Randersacker
  - Nycomed Deutschland GmbH, Ransbach-Baumbach
  - Nycomed Deutschland GmbH, Rastatt
  - Nycomed Deutschland GmbH, Rastede
  - Nycomed Deutschland GmbH, Ratingen
  - Nycomed Deutschland GmbH, Ratzeburg
  - Nycomed Deutschland GmbH, Raubach
  - Nycomed Deutschland GmbH, Raubling
  - Nycomed Deutschland GmbH, Rauenberg
  - Nycomed Deutschland GmbH, Ravensburg
  - Nycomed Deutschland GmbH, Recke
  - Nycomed Deutschland GmbH, Recklinghausen
  - Nycomed Deutschland GmbH, Redefin
  - Nycomed Deutschland GmbH, Redwitz a.d.Rodach
  - Nycomed Deutschland GmbH, Rees
  - Nycomed Deutschland GmbH, Regen
  - Nycomed Deutschland GmbH, Regensburg
  - Nycomed Deutschland GmbH, Regis-Breitingen
  - Nycomed Deutschland GmbH, Rehden
  - Nycomed Deutschland GmbH, Rehlingen-Siersburg
  - Nycomed Deutschland GmbH, Rehna
  - Nycomed Deutschland GmbH, Reichardtswerben
  - Nycomed Deutschland GmbH, Reichenbach
  - Nycomed Deutschland GmbH, Reilingen
  - Nycomed Deutschland GmbH, Reinbek
  - Nycomed Deutschland GmbH, Reinfeld
  - Nycomed Deutschland GmbH, Reinheim
  - Nycomed Deutschland GmbH, Reisbach
  - Nycomed Deutschland GmbH, Reischach
  - Nycomed Deutschland GmbH, Rellingen
  - Nycomed Deutschland GmbH, Remagen
  - Nycomed Deutschland GmbH, Remscheid
  - Nycomed Deutschland GmbH, Renchen
  - Nycomed Deutschland GmbH, Rendsburg
  - Nycomed Deutschland GmbH, Reutlingen
  - Nycomed Deutschland GmbH, Rhaunen
  - Nycomed Deutschland GmbH, Rheinau
  - Nycomed Deutschland GmbH, Rheinbach
  - Nycomed Deutschland GmbH, Rheinberg
  - Nycomed Deutschland GmbH, Rheinbreitbach
  - Nycomed Deutschland GmbH, Rheine
  - Nycomed Deutschland GmbH, Rheinmünster
  - Nycomed Deutschland GmbH, Rheinzabern
  - Nycomed Deutschland GmbH, Rheurdt
  - Nycomed Deutschland GmbH, Rhumspringe
  - Nycomed Deutschland GmbH, Rickenbach
  - Nycomed Deutschland GmbH, Riede
  - Nycomed Deutschland GmbH, Rieden
  - Nycomed Deutschland GmbH, Riegel
  - Nycomed Deutschland GmbH, Riegelsberg
  - Nycomed Deutschland GmbH, Riesa
  - Nycomed Deutschland GmbH, Rietberg
  - Nycomed Deutschland GmbH, Rietz Neuendorf
  - Nycomed Deutschland GmbH, Ringstedt
  - Nycomed Deutschland GmbH, Rinteln
  - Nycomed Deutschland GmbH, Rochlitz
  - Nycomed Deutschland GmbH, Rodalben
  - Nycomed Deutschland GmbH, Rodenbach
  - Nycomed Deutschland GmbH, Roding
  - Nycomed Deutschland GmbH, Roggendorf
  - Nycomed Deutschland GmbH, Rosenheim
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Rotenburg (Wümme)
  - Nycomed Deutschland GmbH, Roxheim
  - Nycomed Deutschland GmbH, Roßbach
  - Nycomed Deutschland GmbH, Rödermark
  - Nycomed Deutschland GmbH, Rödersheim-Gronau
  - Nycomed Deutschland GmbH, Röhrmoos
  - Nycomed Deutschland GmbH, Römerberg
  - Nycomed Deutschland GmbH, Römerstein
  - Nycomed Deutschland GmbH, Rötha
  - Nycomed Deutschland GmbH, Röthenbach a.d.Pegnitz
  - Nycomed Deutschland GmbH, Rudersberg
  - Nycomed Deutschland GmbH, Ruderting
  - Nycomed Deutschland GmbH, Ruhmannsfelden
  - Nycomed Deutschland GmbH, Ruppichteroth
  - Nycomed Deutschland GmbH, Rutesheim
  - Nycomed Deutschland GmbH, Rühen
  - Nycomed Deutschland GmbH, Rülzheim
  - Nycomed Deutschland GmbH, Saal a.d.Donau
  - Nycomed Deutschland GmbH, Saalburg-Ebersdorf
  - Nycomed Deutschland GmbH, Saarbrücken
  - Nycomed Deutschland GmbH, Saarlouis
  - Nycomed Deutschland GmbH, Sachsenheim
  - Nycomed Deutschland GmbH, Saerbeck
  - Nycomed Deutschland GmbH, Saint Blasien
  - Nycomed Deutschland GmbH, Saint Georgen Im Schwarzwald
  - Nycomed Deutschland GmbH, Saint Johann
  - Nycomed Deutschland GmbH, Saint Wendel
  - Nycomed Deutschland GmbH, Salem
  - Nycomed Deutschland GmbH, Salzgitter
  - Nycomed Deutschland GmbH, Salzkotten
  - Nycomed Deutschland GmbH, Salzmünde
  - Nycomed Deutschland GmbH, Salzwedel
  - Nycomed Deutschland GmbH, Sand A. Main
  - Nycomed Deutschland GmbH, Sande
  - Nycomed Deutschland GmbH, Sandersdorf
  - Nycomed Deutschland GmbH, Sandesneben
  - Nycomed Deutschland GmbH, Sandhausen
  - Nycomed Deutschland GmbH, Sangerhausen
  - Nycomed Deutschland GmbH, Sankt Goar
  - Nycomed Deutschland GmbH, Sassnitz
  - Nycomed Deutschland GmbH, Saterland
  - Nycomed Deutschland GmbH, Saubach
  - Nycomed Deutschland GmbH, Schalkau
  - Nycomed Deutschland GmbH, Schalksmühle
  - Nycomed Deutschland GmbH, Schellerten
  - Nycomed Deutschland GmbH, Schenefeld
  - Nycomed Deutschland GmbH, Scheßlitz
  - Nycomed Deutschland GmbH, Schiffdorf
  - Nycomed Deutschland GmbH, Schifferstadt
  - Nycomed Deutschland GmbH, Schiffweiler
  - Nycomed Deutschland GmbH, Schillsdorf
  - Nycomed Deutschland GmbH, Schirnding
  - Nycomed Deutschland GmbH, Schkeuditz
  - Nycomed Deutschland GmbH, Schleching
  - Nycomed Deutschland GmbH, Schlehdorf
  - Nycomed Deutschland GmbH, Schleiz
  - Nycomed Deutschland GmbH, Schleusingen
  - Nycomed Deutschland GmbH, Schmalkalden
  - Nycomed Deutschland GmbH, Schmallenberg
  - Nycomed Deutschland GmbH, Schmidmühlen
  - Nycomed Deutschland GmbH, Schmiedeberg
  - Nycomed Deutschland GmbH, Schmölln-Putzkau
  - Nycomed Deutschland GmbH, Schnaittach
  - Nycomed Deutschland GmbH, Schneeberg
  - Nycomed Deutschland GmbH, Schongau
  - Nycomed Deutschland GmbH, Schopfloch
  - Nycomed Deutschland GmbH, Schorndorf
  - Nycomed Deutschland GmbH, Schönberg
  - Nycomed Deutschland GmbH, Schönebeck
  - Nycomed Deutschland GmbH, Schönefeld
  - Nycomed Deutschland GmbH, Schönenberg-Kübelberg
  - Nycomed Deutschland GmbH, Schönfeld
  - Nycomed Deutschland GmbH, Schönsee
  - Nycomed Deutschland GmbH, Schönwalde-Glien
  - Nycomed Deutschland GmbH, Schöppenstedt
  - Nycomed Deutschland GmbH, Schramberg
  - Nycomed Deutschland GmbH, Schriesheim
  - Nycomed Deutschland GmbH, Schutterwald
  - Nycomed Deutschland GmbH, Schwabach
  - Nycomed Deutschland GmbH, Schwabmünchen
  - Nycomed Deutschland GmbH, Schwaikheim
  - Nycomed Deutschland GmbH, Schwalbach am Taunus
  - Nycomed Deutschland GmbH, Schwalmstadt
  - Nycomed Deutschland GmbH, Schwanau
  - Nycomed Deutschland GmbH, Schwandorf in Bayern
  - Nycomed Deutschland GmbH, Schwanewede
  - Nycomed Deutschland GmbH, Schwangau
  - Nycomed Deutschland GmbH, Schwarmstedt
  - Nycomed Deutschland GmbH, Schwarz
  - Nycomed Deutschland GmbH, Schwarza
  - Nycomed Deutschland GmbH, Schwarzach
  - Nycomed Deutschland GmbH, Schwarzenbach A Wald
  - Nycomed Deutschland GmbH, Schwarzheide
  - Nycomed Deutschland GmbH, Schwäbisch Gmünd
  - Nycomed Deutschland GmbH, Schwedt
  - Nycomed Deutschland GmbH, Schweich
  - Nycomed Deutschland GmbH, Schweinfurt
  - Nycomed Deutschland GmbH, Schwelm
  - Nycomed Deutschland GmbH, Schwentinental
  - Nycomed Deutschland GmbH, Schwerin
  - Nycomed Deutschland GmbH, Schwerte
  - Nycomed Deutschland GmbH, Schwetzingen
  - Nycomed Deutschland GmbH, Seehausen
  - Nycomed Deutschland GmbH, Seelow
  - Nycomed Deutschland GmbH, Seesen
  - Nycomed Deutschland GmbH, Sehnde
  - Nycomed Deutschland GmbH, Selsingen
  - Nycomed Deutschland GmbH, Selters
  - Nycomed Deutschland GmbH, Senden
  - Nycomed Deutschland GmbH, Seubersdorf i.d.OPf.
  - Nycomed Deutschland GmbH, Siegen
  - Nycomed Deutschland GmbH, Siegsdorf
  - Nycomed Deutschland GmbH, Sievershagen
  - Nycomed Deutschland GmbH, Sigmaringen
  - Nycomed Deutschland GmbH, Silberhausen
  - Nycomed Deutschland GmbH, Silberstedt
  - Nycomed Deutschland GmbH, Sindelfingen
  - Nycomed Deutschland GmbH, Singen
  - Nycomed Deutschland GmbH, Sinsheim
  - Nycomed Deutschland GmbH, Sinzing
  - Nycomed Deutschland GmbH, Solingen
  - Nycomed Deutschland GmbH, Solms
  - Nycomed Deutschland GmbH, Soltau
  - Nycomed Deutschland GmbH, Sondershausen
  - Nycomed Deutschland GmbH, Sonneberg
  - Nycomed Deutschland GmbH, Sonthofen
  - Nycomed Deutschland GmbH, Sontra
  - Nycomed Deutschland GmbH, Söhrewald
  - Nycomed Deutschland GmbH, Sömmerda
  - Nycomed Deutschland GmbH, Spalt
  - Nycomed Deutschland GmbH, Spardorf
  - Nycomed Deutschland GmbH, Spechbach
  - Nycomed Deutschland GmbH, Speicher
  - Nycomed Deutschland GmbH, Speichersdorf
  - Nycomed Deutschland GmbH, Spenge
  - Nycomed Deutschland GmbH, Speyer
  - Nycomed Deutschland GmbH, Spiesen-Elversberg
  - Nycomed Deutschland GmbH, Spremberg
  - Nycomed Deutschland GmbH, Sprendlingen
  - Nycomed Deutschland GmbH, Springe
  - Nycomed Deutschland GmbH, Sprockhövel
  - Nycomed Deutschland GmbH, Stade
  - Nycomed Deutschland GmbH, Stadland
  - Nycomed Deutschland GmbH, Stadtbergen
  - Nycomed Deutschland GmbH, Stadtlohn
  - Nycomed Deutschland GmbH, Stadtroda
  - Nycomed Deutschland GmbH, Stahnsdorf
  - Nycomed Deutschland GmbH, Stamsried
  - Nycomed Deutschland GmbH, Staudernheim
  - Nycomed Deutschland GmbH, Staßfurt
  - Nycomed Deutschland GmbH, Steigra
  - Nycomed Deutschland GmbH, Steinach
  - Nycomed Deutschland GmbH, Steinen
  - Nycomed Deutschland GmbH, Steinfurt
  - Nycomed Deutschland GmbH, Steinhagen
  - Nycomed Deutschland GmbH, Steinwiesen
  - Nycomed Deutschland GmbH, Steißlingen
  - Nycomed Deutschland GmbH, Stemwede
  - Nycomed Deutschland GmbH, Stendal
  - Nycomed Deutschland GmbH, Sternberg
  - Nycomed Deutschland GmbH, Stockelsdorf
  - Nycomed Deutschland GmbH, Stolberg
  - Nycomed Deutschland GmbH, Stollberg
  - Nycomed Deutschland GmbH, Stolpen
  - Nycomed Deutschland GmbH, Stralsund
  - Nycomed Deutschland GmbH, Straubing
  - Nycomed Deutschland GmbH, Strausberg
  - Nycomed Deutschland GmbH, Straßkirchen
  - Nycomed Deutschland GmbH, Striegistal
  - Nycomed Deutschland GmbH, Stuhr
  - Nycomed Deutschland GmbH, Stuttgart
  - Nycomed Deutschland GmbH, Stützengrün
  - Nycomed Deutschland GmbH, Suhl
  - Nycomed Deutschland GmbH, Sulingen
  - Nycomed Deutschland GmbH, Sulz am Neckar
  - Nycomed Deutschland GmbH, Sulzbach
  - Nycomed Deutschland GmbH, Sulzbach A. Main
  - Nycomed Deutschland GmbH, Sulzbach-Rosenberg
  - Nycomed Deutschland GmbH, Sulzheim
  - Nycomed Deutschland GmbH, Surwold
  - Nycomed Deutschland GmbH, Südharz
  - Nycomed Deutschland GmbH, Sünching
  - Nycomed Deutschland GmbH, Taarstedt
  - Nycomed Deutschland GmbH, Tamm
  - Nycomed Deutschland GmbH, Tangerhütte
  - Nycomed Deutschland GmbH, Tann
  - Nycomed Deutschland GmbH, Tanna
  - Nycomed Deutschland GmbH, Taucha
  - Nycomed Deutschland GmbH, Tauche
  - Nycomed Deutschland GmbH, Teltow
  - Nycomed Deutschland GmbH, Templin
  - Nycomed Deutschland GmbH, Tengen
  - Nycomed Deutschland GmbH, Teningen
  - Nycomed Deutschland GmbH, Teterow
  - Nycomed Deutschland GmbH, Tettnang
  - Nycomed Deutschland GmbH, Teublitz
  - Nycomed Deutschland GmbH, Teuchern
  - Nycomed Deutschland GmbH, Thaleischweiler-Fröschen
  - Nycomed Deutschland GmbH, Thedinghausen
  - Nycomed Deutschland GmbH, Themar
  - Nycomed Deutschland GmbH, Timmendorfer Strand
  - Nycomed Deutschland GmbH, Titisee-Neustadt
  - Nycomed Deutschland GmbH, Tittmoning
  - Nycomed Deutschland GmbH, Todtmoos
  - Nycomed Deutschland GmbH, Torgau
  - Nycomed Deutschland GmbH, Torgelow
  - Nycomed Deutschland GmbH, Tostedt
  - Nycomed Deutschland GmbH, Töging A. Inn
  - Nycomed Deutschland GmbH, Tönisvorst
  - Nycomed Deutschland GmbH, Trappenkamp
  - Nycomed Deutschland GmbH, Traunreut
  - Nycomed Deutschland GmbH, Treffurt
  - Nycomed Deutschland GmbH, Treis-Karden
  - Nycomed Deutschland GmbH, Treuchtlingen
  - Nycomed Deutschland GmbH, Treuen
  - Nycomed Deutschland GmbH, Treuenbrietzen
  - Nycomed Deutschland GmbH, Tribsees
  - Nycomed Deutschland GmbH, Trier
  - Nycomed Deutschland GmbH, Triptis
  - Nycomed Deutschland GmbH, Trittau
  - Nycomed Deutschland GmbH, Troisdorf
  - Nycomed Deutschland GmbH, Trossingen
  - Nycomed Deutschland GmbH, Trostberg an der Alz
  - Nycomed Deutschland GmbH, Türkheim
  - Nycomed Deutschland GmbH, Ubstadt-Weiher
  - Nycomed Deutschland GmbH, Uder
  - Nycomed Deutschland GmbH, Ueckermünde
  - Nycomed Deutschland GmbH, Uelsen
  - Nycomed Deutschland GmbH, Uelzen
  - Nycomed Deutschland GmbH, Uetersen
  - Nycomed Deutschland GmbH, Uettingen
  - Nycomed Deutschland GmbH, Ulm
  - Nycomed Deutschland GmbH, Unna
  - Nycomed Deutschland GmbH, Unterbreizbach
  - Nycomed Deutschland GmbH, Unterföhring
  - Nycomed Deutschland GmbH, Unterhaching
  - Nycomed Deutschland GmbH, Unterkirnach
  - Nycomed Deutschland GmbH, Unterneukirchen
  - Nycomed Deutschland GmbH, Unterpleichfeld
  - Nycomed Deutschland GmbH, Unterschneidheim
  - Nycomed Deutschland GmbH, Untershausen
  - Nycomed Deutschland GmbH, Unterwellenborn
  - Nycomed Deutschland GmbH, Urbach
  - Nycomed Deutschland GmbH, Urspringen
  - Nycomed Deutschland GmbH, Übach-Palenberg
  - Nycomed Deutschland GmbH, Vachendorf
  - Nycomed Deutschland GmbH, Vallendar
  - Nycomed Deutschland GmbH, Varel
  - Nycomed Deutschland GmbH, Vechelde
  - Nycomed Deutschland GmbH, Vechta
  - Nycomed Deutschland GmbH, Veilsdorf
  - Nycomed Deutschland GmbH, Veitsbronn
  - Nycomed Deutschland GmbH, Velbert
  - Nycomed Deutschland GmbH, Velburg
  - Nycomed Deutschland GmbH, Velden
  - Nycomed Deutschland GmbH, Vellahn
  - Nycomed Deutschland GmbH, Vellmar
  - Nycomed Deutschland GmbH, Velten
  - Nycomed Deutschland GmbH, Verden an der Aller
  - Nycomed Deutschland GmbH, Veringenstadt
  - Nycomed Deutschland GmbH, Vetschau
  - Nycomed Deutschland GmbH, Viersen
  - Nycomed Deutschland GmbH, Villingen-Schwenningen
  - Nycomed Deutschland GmbH, Vilshofen
  - Nycomed Deutschland GmbH, Voerde
  - Nycomed Deutschland GmbH, Vogtsburg
  - Nycomed Deutschland GmbH, Vöhrenbach
  - Nycomed Deutschland GmbH, Vöhringen
  - Nycomed Deutschland GmbH, Völkershausen
  - Nycomed Deutschland GmbH, Völklingen
  - Nycomed Deutschland GmbH, Waakirchen
  - Nycomed Deutschland GmbH, Wachtendonk
  - Nycomed Deutschland GmbH, Wadgassen
  - Nycomed Deutschland GmbH, Wagenfeld
  - Nycomed Deutschland GmbH, Waiblingen
  - Nycomed Deutschland GmbH, Waidhaus
  - Nycomed Deutschland GmbH, Waldalgesheim
  - Nycomed Deutschland GmbH, Waldaschaff
  - Nycomed Deutschland GmbH, Waldbreitbach
  - Nycomed Deutschland GmbH, Waldenbuch
  - Nycomed Deutschland GmbH, Waldfeucht
  - Nycomed Deutschland GmbH, Waldfischbach-Burgalben
  - Nycomed Deutschland GmbH, Waldheim
  - Nycomed Deutschland GmbH, Waldkirch
  - Nycomed Deutschland GmbH, Waldkraiburg
  - Nycomed Deutschland GmbH, Waldmünchen
  - Nycomed Deutschland GmbH, Wallenhorst
  - Nycomed Deutschland GmbH, Wallerfing
  - Nycomed Deutschland GmbH, Wallgau
  - Nycomed Deutschland GmbH, Wallhausen
  - Nycomed Deutschland GmbH, Wallmerod
  - Nycomed Deutschland GmbH, Walsrode
  - Nycomed Deutschland GmbH, Walzbachtal
  - Nycomed Deutschland GmbH, Wanfried
  - Nycomed Deutschland GmbH, Wangen
  - Nycomed Deutschland GmbH, Wangerland
  - Nycomed Deutschland GmbH, Wankendorf
  - Nycomed Deutschland GmbH, Wanzleben-Börde
  - Nycomed Deutschland GmbH, Warburg
  - Nycomed Deutschland GmbH, Warin
  - Nycomed Deutschland GmbH, Warnow
  - Nycomed Deutschland GmbH, Warstein
  - Nycomed Deutschland GmbH, Warthausen
  - Nycomed Deutschland GmbH, Wassenberg
  - Nycomed Deutschland GmbH, Wattenheim
  - Nycomed Deutschland GmbH, Wedel
  - Nycomed Deutschland GmbH, Weeze
  - Nycomed Deutschland GmbH, Wegberg
  - Nycomed Deutschland GmbH, Weibern
  - Nycomed Deutschland GmbH, Weida
  - Nycomed Deutschland GmbH, Weiden i.d.OPf.
  - Nycomed Deutschland GmbH, Weil am Rhein
  - Nycomed Deutschland GmbH, Weilburg
  - Nycomed Deutschland GmbH, Weilerswist
  - Nycomed Deutschland GmbH, Weilheim an der Teck
  - Nycomed Deutschland GmbH, Weilheim I. OB
  - Nycomed Deutschland GmbH, Weinbergen
  - Nycomed Deutschland GmbH, Weingarten
  - Nycomed Deutschland GmbH, Weinheim
  - Nycomed Deutschland GmbH, Weinsberg
  - Nycomed Deutschland GmbH, Weinstadt
  - Nycomed Deutschland GmbH, Weiskirchen
  - Nycomed Deutschland GmbH, Weissensee
  - Nycomed Deutschland GmbH, Weitramsdorf
  - Nycomed Deutschland GmbH, Weißach
  - Nycomed Deutschland GmbH, Weißandt-Gölzau
  - Nycomed Deutschland GmbH, Weißenfels
  - Nycomed Deutschland GmbH, Weißenhorn
  - Nycomed Deutschland GmbH, Weißenthurm
  - Nycomed Deutschland GmbH, Weißwasser
  - Nycomed Deutschland GmbH, Welden
  - Nycomed Deutschland GmbH, Welver
  - Nycomed Deutschland GmbH, Welzheim
  - Nycomed Deutschland GmbH, Wendeburg
  - Nycomed Deutschland GmbH, Wendelstein
  - Nycomed Deutschland GmbH, Wennigsen
  - Nycomed Deutschland GmbH, Werdau
  - Nycomed Deutschland GmbH, Werder
  - Nycomed Deutschland GmbH, Werne
  - Nycomed Deutschland GmbH, Werneck
  - Nycomed Deutschland GmbH, Werneuchen
  - Nycomed Deutschland GmbH, Wernigerode
  - Nycomed Deutschland GmbH, Wertheim am Main
  - Nycomed Deutschland GmbH, Wesel
  - Nycomed Deutschland GmbH, Wesselburen
  - Nycomed Deutschland GmbH, Wesseling
  - Nycomed Deutschland GmbH, Westerburg
  - Nycomed Deutschland GmbH, Westerkappeln
  - Nycomed Deutschland GmbH, Westerland
  - Nycomed Deutschland GmbH, Westerstede
  - Nycomed Deutschland GmbH, Westoverledingen
  - Nycomed Deutschland GmbH, Wettenberg
  - Nycomed Deutschland GmbH, Wetter
  - Nycomed Deutschland GmbH, Wetterzeube
  - Nycomed Deutschland GmbH, Wettin
  - Nycomed Deutschland GmbH, Wetzlar
  - Nycomed Deutschland GmbH, Weyerbusch
  - Nycomed Deutschland GmbH, Weyhe
  - Nycomed Deutschland GmbH, Wickede
  - Nycomed Deutschland GmbH, Wiehl
  - Nycomed Deutschland GmbH, Wiesbaden
  - Nycomed Deutschland GmbH, Wiesenfelden
  - Nycomed Deutschland GmbH, Wiesloch
  - Nycomed Deutschland GmbH, Wietmarschen
  - Nycomed Deutschland GmbH, Wietzen
  - Nycomed Deutschland GmbH, Wiggensbach
  - Nycomed Deutschland GmbH, Wilburgstetten
  - Nycomed Deutschland GmbH, Wildenfels
  - Nycomed Deutschland GmbH, Wildeshausen
  - Nycomed Deutschland GmbH, Wilhelmshaven
  - Nycomed Deutschland GmbH, Wilkau-Haßlau
  - Nycomed Deutschland GmbH, Willebadessen
  - Nycomed Deutschland GmbH, Willich
  - Nycomed Deutschland GmbH, Wilster
  - Nycomed Deutschland GmbH, Wilthen
  - Nycomed Deutschland GmbH, Winhöring
  - Nycomed Deutschland GmbH, Winnenden
  - Nycomed Deutschland GmbH, Winsen
  - Nycomed Deutschland GmbH, Winterberg
  - Nycomed Deutschland GmbH, Winterstein
  - Nycomed Deutschland GmbH, Wismar
  - Nycomed Deutschland GmbH, Witten
  - Nycomed Deutschland GmbH, Wittenberg
  - Nycomed Deutschland GmbH, Wittenberge
  - Nycomed Deutschland GmbH, Wittenburg
  - Nycomed Deutschland GmbH, Wittgensdorf
  - Nycomed Deutschland GmbH, Wittlich
  - Nycomed Deutschland GmbH, Wittstock
  - Nycomed Deutschland GmbH, Witzenhausen
  - Nycomed Deutschland GmbH, Wolfach
  - Nycomed Deutschland GmbH, Wolfenbüttel
  - Nycomed Deutschland GmbH, Wolfratshausen
  - Nycomed Deutschland GmbH, Wolfsberg
  - Nycomed Deutschland GmbH, Wolfsburg
  - Nycomed Deutschland GmbH, Wollin
  - Nycomed Deutschland GmbH, Wolnzach
  - Nycomed Deutschland GmbH, Woltersdorf
  - Nycomed Deutschland GmbH, Worbis
  - Nycomed Deutschland GmbH, Worms
  - Nycomed Deutschland GmbH, Wormstedt
  - Nycomed Deutschland GmbH, Wotenitz
  - Nycomed Deutschland GmbH, Wölfersheim
  - Nycomed Deutschland GmbH, Wörrstadt
  - Nycomed Deutschland GmbH, Wörth a.d.Donau
  - Nycomed Deutschland GmbH, Wörth am Rhein
  - Nycomed Deutschland GmbH, Wriedel
  - Nycomed Deutschland GmbH, Wriezen
  - Nycomed Deutschland GmbH, Wrist
  - Nycomed Deutschland GmbH, Wunstorf
  - Nycomed Deutschland GmbH, Wuppertal
  - Nycomed Deutschland GmbH, Wurmberg
  - Nycomed Deutschland GmbH, Wurzen
  - Nycomed Deutschland GmbH, Wustermark
  - Nycomed Deutschland GmbH, Wutha
  - Nycomed Deutschland GmbH, Würselen
  - Nycomed Deutschland GmbH, Würzburg
  - Nycomed Deutschland GmbH, Zapfendorf
  - Nycomed Deutschland GmbH, Zehdenick
  - Nycomed Deutschland GmbH, Zeitz
  - Nycomed Deutschland GmbH, Zell
  - Nycomed Deutschland GmbH, Zell unter Aichelberg
  - Nycomed Deutschland GmbH, Zerbst
  - Nycomed Deutschland GmbH, Zernitz-Lohm
  - Nycomed Deutschland GmbH, Zeschendorf
  - Nycomed Deutschland GmbH, Zetel
  - Nycomed Deutschland GmbH, Zeulenroda-Triebes
  - Nycomed Deutschland GmbH, Zirndorf
  - Nycomed Deutschland GmbH, Zittau
  - Nycomed Deutschland GmbH, Zorge
  - Nycomed Deutschland GmbH, Zörbig
  - Nycomed Deutschland GmbH, Zschopau
  - Nycomed Deutschland GmbH, Zschornewitz
  - Nycomed Deutschland GmbH, Zwenkau
  - Nycomed Deutschland GmbH, Zwickau
  - Nycomed Deutschland GmbH, Zwiesel
  - Nycomed Deutschland GmbH, Zwota
  - Nycomed Deutschland GmbH, Zwönitz